CLINICAL TRIAL: NCT02200263
Title: A Randomized Placebo-controlled Trial to Investigate the Effect of Lutein and Zeaxanthin Supplementation on Macular Pigment and Visual Function in Albinism - LUtein for VIsion in Albinism (LUVIA)
Brief Title: The Effects of Lutein and Zeaxanthin Supplementation on Vision in Patients With Albinism
Acronym: LUVIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Clark Charitable Foundation Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA_00088335
Record Dates: First submitted 2014-07-23; First posted 2014-07-25 (Estimated); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Ocular Albinism (OA); Oculocutaneous Albinism (OCA)
Keywords: ocular albinism (OA); oculocutaneous albinism (OCA); macular pigment; visual function
MeSH Terms: conditions — Albinism, Ocular; Albinism, Oculocutaneous | interventions — Lutein; Zeaxanthins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lutein plus Zeaxanthin (Experimental): Participants randomized to this arm will receive 20 mg of Lutein (L) plus 20 mg of Zeaxanthin (Z) per day: Two pills (10 mg L+ 10 mg Z per pill) for the duration of one year.
  Interventions: Dietary Supplement: Lutein plus Zeaxanthin
- Placebo softgels (Placebo Comparator): Participants randomized to this arm will receive two pills per day of placebo-gels corresponding to the active compound in look and feel for the duration of one year
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lutein plus Zeaxanthin — dose: two softgels once a day with a meal
  Other Names: EyePromise® Lutein + Zeaxanthin (ZeaVision, LLC)
  Arms: Lutein plus Zeaxanthin
Dietary Supplement: Placebo — two softgels once-daily with a meal
  Other Names: placebo softgels
  Arms: Placebo softgels

SUMMARY:
The LUVIA study is a randomized placebo-controlled trial designed to investigate the effects of lutein and zeaxanthin supplementation on macular pigment and visual function in ocular or oculocutaneous albinism. Lutein and zeaxanthin supplementation will be compared to a placebo (no treatment) gel pill over the period of 12 months, with study visits approximately every 3 months for the first year and a final visit 18 months after enrollment.

DETAILED DESCRIPTION:
Ocular and oculocutaneous albinism represent a spectrum of disorders with absent or significantly diminished amount of melanin either across different body tissues - skin, hair, eye (Oculocutaneous Albinism 1 and 2), or exclusively in eye tissues only (Ocular Albinism 1) .

The functionality and the clinical findings are diverse (the phenotype), and no direct correlation has been established to the underlying mutations (genotype).

The common ocular phenotype includes iris transillumination, foveal hypoplasia, nystagmus, reduced visual acuity, refractive error, photosensitivity and abnormal development of the visual pathways with characteristic abnormal routing of ganglion cell axons in the chiasma, resulting in abnormal visually evoked potentials. Current treatment options are limited to optical methods and low vision aids.

The mechanism of melanin pigment formation in the RPE cells and its role in the visual pathways and structures development is not completely understood, but a correlation was found between the amount of fundus pigmentation and visual function in albino patients. The absent pigmentation within the retinal pigment epithelium (RPE) may thus contribute to visual performance deficits.

The macular pigment (MP) consists of two main carotenoids, lutein and zeaxanthin, which are concentrated in the macular region of the retina. MP is hypothesized to function via a protective mechanism by absorbing blue light incident on the retina thereby reducing oxidative damage to the underlying photoreceptors. It is also thought to improve visual function via reduction of chromatic aberration and glare. It is currently unclear as to how the variability in macular pigment optical density (MPOD) affects congenital retinal conditions. The MP would, however, be a hypothetical and good candidate to improve visual performance - simply by increasing pigmentation, reducing light scatter and thus glare sensitivity.

As this pigment is not produced in the retina, but is absorbed via diet, it can be manipulated by alteration in diet and supplementation thereby providing potential therapy for retinal diseases. It is however necessary first to see if MPOD levels are measurable in this disorder before dietary advice can be provided after completion of the LUVIA study. Further to this, evaluation of both the structural and functional properties of the retina will provide greater insight into the possible function of MP in this retinal disease including whether supplementation would be of benefit.

ELIGIBILITY:
Inclusion Criteria:

* Age of 12 years old and older
* Clinical and/or genetic diagnosis of ocular or oculocutaneous albinism
* Ocular media allowing acceptable visualization of the retina.
* Ocular media allowing acceptable quality of the ocular coherence tomography (OCT) and/or fundus autofluorescence (FAF) scans.
* At least one reliable central macular pigment optical density (MPOD) measurement captured on the enrollment visit in at least one eligible eye
* Best corrected visual acuity of 20/200 or better in one or both eligible eyes (eyes that confirmed to be eligible by the MPOD testing).

Exclusion Criteria:

* Persons taking lutein and/or zeaxanthin supplements over the past 6 months
* Pregnant or planning to become pregnant
* Evidence of present or past retinal macular condition other than congenital foveal hypoplasia
* History of gastrointestinal disease that would interfere with absorption of lutein and zeaxanthin
* Participation in a clinical trial requiring visual testing or administration of a drug (marketed or investigational) within 60 days before entry in the study (the day informed consent is signed)
* Inability to communicate or cooperate with the investigator due to cognitive impairment or poor general health
* Any other condition which, in the opinion of the investigators, is likely to interfere with the successful collection of the measures required for the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Macular pigment optical density (MPOD) | 12 months
  MPOD will be measured at baseline and follow-up. MPOD will be evaluated psychophysically using the QuantifEye device (ZeaVision), optically using the MPOD module of the Heidelberg Spectralis multicolor imaging device, and by quantitative fundus autofluorescence (FAF) using the Heidelberg Spectralis multicolor imaging device

SECONDARY OUTCOMES:
Contrast acuity | 12 months
  Contrast acuity will be measured at baseline and follow-up using the Innova electronic visual system and the quick Contrast Sensitivity Function (Adaptive Sensory Technology, LLC)
Visual field, fixation and central retinal sensitivity | 12 months
  Microperimetry testing via the microperimetry (MP) -1 device (Nidek) will be performed at baseline and follow-up
Bioavailability profile of Lutein and Zeaxanthin | 12 months
  Blood samples will be collected at follow-up, and Lutein and Zeaxanthin concentration levels assessed.
Evaluation of the diversity of microstructural central retinal abnormalities | 12 months
  Spectral domain ocular coherence tomography (SD-OCT) macular scan will be performed at baseline and at 12 months
Best Corrected Visual Acuity (BCVA) | 12 months
  BCVA will evaluated using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol at baseline and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Neil Bressler, MD, Principal Investigator — Johns Hopkins University; Mary E. Frey, Study Director — Johns Hopkins University
Locations (1):
- Wilmer Eye Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No